CLINICAL TRIAL: NCT00123331
Title: Rapamycin Use in CNI-Free Immunosuppression for Stabilization/Improvement of Renal Function After Heart Transplantation
Brief Title: Rapamycin Use in Calcineurin Inhibitor (CNI)-Free Immunosuppression for Stabilization/Improvement of Renal Function After Heart Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD_cardio_352/2003_dengler
Record Dates: First submitted 2005-07-18; First posted 2005-07-22 (Estimated); Last update posted 2005-08-02 (Estimated); Status verified 2005-06

CONDITIONS: Heart Transplantation; Renal Failure
Keywords: Heart transplantation; Renal failure; Cyclosporine; Rapamycin
MeSH Terms: conditions — Renal Insufficiency

INTERVENTIONS:
Drug: Cyclosporine discontinuation
Drug: Rapamycin medication

SUMMARY:
Clinical Problem: Renal insufficiency after heart transplantation caused by cyclosporine medication was addressed. Current therapeutic approaches include cyclosporine reduction or discontinuation. It is unclear whether discontinuation of low dose cyclosporine also has a beneficial effect, i.e. is there a threshold effect for cyclosporine nephrotoxicity?

Study Design: Heart transplant patients with a moderate degree of renal failure on low dose cyclosporine were randomized to either a) no change; or b) discontinuation of cyclosporine and initiation of rapamycin immunosuppression.

Read-Out: Renal function after 6 months; tolerability; and safety were assessed.

DETAILED DESCRIPTION:
Clinical Problem: Renal insufficiency after heart transplantation caused by cyclosporine medication was addressed. Current therapeutic approaches include cyclosporine reduction or discontinuation. It is unclear whether discontinuation of low dose cyclosporine also has a beneficial effect, i.e. is there a threshold effect for cyclosporine nephrotoxicity?

Study Design: Heart transplant patients with a moderate degree of renal failure on low dose cyclosporine were randomized to either a) no change; or b) discontinuation of cyclosporine and initiation of rapamycin immunosuppression.

Read-Out: Renal function after 6 months; tolerability; and safety were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplantation (> 6 months post-operation)
* Renal failure (serum creatinine stably > 1.7 mg/dl
* Cyclosporine trough blood level < 110 ng/ml

Exclusion Criteria:

* < 18 years of age
* Rapamycin intolerability
* Active infection
* Pregnancy, breast feeding
* Major elective surgery planned in study period
* Thrombopenia < 100,000/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Study Completion 2005-04

PRIMARY OUTCOMES:
Renal function after 6 months (serum creatinine, calculated creatinine clearance)

SECONDARY OUTCOMES:
Survival
Rejection (clinical)
Tolerability
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Dengler, MD, Principal Investigator — Heidelberg University
Locations (1):
- Medizinische Universitätsklinik, Kardiologie, Heidelberg, Germany

REFERENCES:
- [Background] Angermann CE, Stork S, Costard-Jackle A, Dengler TJ, Siebert U, Tenderich G, Rahmel A, Schwarz ER, Nagele H, Wagner FM, Haaff B, Pethig K. Reduction of cyclosporine after introduction of mycophenolate mofetil improves chronic renal dysfunction in heart transplant recipients--the IMPROVED multi-centre study. Eur Heart J. 2004 Sep;25(18):1626-34. doi: 10.1016/j.ehj.2004.06.032. PMID 15351162